CLINICAL TRIAL: NCT05678270
Title: A Single-Arm, Open-Label, Multicenter Phase II Study to Evaluate the Efficacy and Safety of ICP-192 in Subjects With Unresectable or Metastatic Intrahepatic Cholangiocarcinoma With FGFR2 Fusions/Rearrangements Who Have Failed Prior Therapy
Brief Title: A Study of ICP-192 in Patients With FGFR2-Rearranged Unresectable or Metastatic Intrahepatic Cholangiocarcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Beijing InnoCare Pharma Tech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ICP-CL-00305
Record Dates: First submitted 2022-12-23; First posted 2023-01-10 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Intrahepatic Cholangiocarcinoma (ICC)
MeSH Terms: conditions — Cholangiocarcinoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ICP-192 (Experimental)
  Interventions: Drug: ICP-192

INTERVENTIONS:
Drug: ICP-192 — ICP-192 is a round, uncoated tablet, 5mg, orally.

SUMMARY:
This is a single-arm, open-label, multi-center phase 2 clinical trial of ICP-192. The purpose of this study is to evaluate the efficacy and safety in patients with FGFR2-Rearranged unresectable or metastatic intrahepatic cholangiocarcinoma who failed prior therapy

ELIGIBILITY:
Inclusion Criteria:

1. Signed the ICF and Age ≥ 18 years old, either sex.
2. ECOG score of 0-1.
3. Life expectancy > 3 months.
4. Histopathologically or cytopathologically confirmed intrahepatic cholangiocarcinoma with unresectable, recurrent or metastatic (AJCC 2017, 8th edition, TNM stage IV) tumor that has progressed following at least one line of chemotherapy and progression/recurrence within 6 months after neoadjuvant/adjuvant chemotherapy may be included.
5. FGFR2 fusion /rearrangement as confirmed by the central laboratory.
6. At least one measurable lesion at screening as target lesion per RECIST 1.1.
7. Organ functions meeting the protocol requirements.
8. Contraception according to the protocol requirements.

Exclusion Criteria:

1. Presence of other malignancies requiring medical intervention.
2. Prior treatment with selective FGFR inhibitors or FGFR antibodies.
3. Treatment with biological products, radical radiotherapy, and other investigational drugs within 4 weeks prior to the first dose of study drug. Chemotherapy within 3 weeks prior to the first dose of study drug.
4. Known symptomatic central nervous system (CNS) metastases.
5. Patients who have not recovered from the toxicity caused by previous anti-tumor treatment and have ≥ Grade 2 adverse events (judged per CTCAE V5.0 evaluation criterion) at the first dose of study drug.
6. Currently uncontrolled cardiovascular and cerebrovascular diseases, or a past medical history.
7. Any unstable or uncontrolled systemic disease as judged by the investigator, such as: active infection requiring intravenous therapy, uncontrolled hypertension (After treatment systolic blood pressure ≥ 150 mmHg and/or diastolic blood pressure ≥ 90 mmHg), and diabetes mellitus (HbA1c > 8%).
8. Current active bleeding, such as deep venous thrombosis, portal hypertension signs leading to gastroesophageal venous bleeding.
9. Wound with active infection.
10. Major surgical procedures within 4 weeks prior to the first dose of the study drug or minor surgical procedures within 2 weeks prior to the first dose of the study drug.
11. Any corneal or retinal abnormalities that may result in an increased risk of ocular toxicity
12. History and/or current evidence of extensive tissue calcification, including but not limited to calcification in soft tissues, kidney, intestine, myocardium, vasculature and/or the lungs, with the exception of lymph node calcification, mild pulmonary parenchymal calcification, and asymptomatic coronary artery calcification.
13. Clinically serious gastrointestinal dysfunction that may affect the intake, transport or absorption of the study drug (such as poorly controlled nausea, vomiting, diarrhea; malabsorption syndrome; intestinal obstruction and small bowel resection, etc.), or the patient was unable to swallow the drug orally.
14. Active HBV infection, Active HCV infection, HIV infection.
15. Female subjects who are pregnant or breastfeeding, or plan to have a pregnancy within 6 months after the last dose of the study drug; or male subjects who plan to father a child during the study or within 6 months after the last dose of the study drug.
16. The last dose of strong CYP3A inhibitor or CYP3A inducer (including food, western medicine, traditional Chinese medicine) is less than 5 half-lives before the first dose of study drug, or plans to take concomitant drugs or foods with strong CYP3A inhibition or induction during the study.
17. Known allergy to any excipients of the study drug.
18. Subjects with conditions that in the investigator's opinion are not suitable for participating in this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2022-11-15 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Up to 3 years

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Up to 3 years
Disease control rate (DCR) | Up to 3 years
Duration of response (DOR) | Up to 3 years
Time to response (TTR) | Up to 3 years
Overall survival (OS) | Up to 3 years
The adverse event (AE) of ICP-192 assessed by NCI-CTCAE V5.0 | Up to 3 years
Maximum concentration (Cmax) | Up to 3 years
Time to maximum concentration (Tmax) | Up to 3 years
Half-life (T1/2) | Up to 3 years
Area under the concentration-time curve (AUC) | Up to 3 years
Apparent clearance (CL/F) | Up to 3 years
Terminal apparent volume of distribution (Vz/F) | Up to 3 years

OTHER OUTCOMES:
To explore the relationship between blood phosphorus and clinical efficacy | Up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Jin Li, Principal Investigator — Shanghai East Hospital
Locations (44):
- China (44):
  - Anhui Provincial Hospital, Hefei, Anhui
  - Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Beijing Youan Hosptital,Capital Medical University, Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Beijing Hospital, Beijing, Beijing Municipality
  - Fujian Cancer Hospital, Fujian, Fujian
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Mengchao hepatobiliary Hospital of FuJian Medical university, Fuzhou, Fujian
  - Foshan First People's Hospital, Foshan, Guangdong
  - Sun Yat-sen Memorial Hospital, Guangzhou, Guangdong
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - ZhuJiang Hospital of Southern Medical University, Guangzhou, Guangdong
  - Hebei Medical University Fourth Hospital, Shijiazhuang, Hebei
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Henan Cancer Hospital, Zhengzhou, Henan
  - First Affiliated Hospital of Zhengzhou University., Zhengzhou, Henan
  - Zhongnan Hospital of Wuhan University, Wuhan, Hubei
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Human Provincial People's Hospital, Changsha, Hunan
  - Hunan Cancer Hospital, Changsha, Hunan
  - The Third Xiangya Hospital of Central South Uninversity, Changsha, Hunan
  - Changzhou Tumor Hospital, Changzhou, Jiangsu
  - Jiangyin Renmin Hospital, Jiangyin, Jiangsu
  - The Affiliated Hospital of Nanjing University Meidical School, Nanjing, Jiangsu
  - The Second Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Xuzhou Central Hospital, Xuzhou, Jiangsu
  - The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - Liaoning Cancer Hospital&Institute, Shenyang, Liaoning
  - Jiangxi Cancer Hospital, Nanchang, Nanchang
  - General Hospital of Ningxia Medical University, Yinchuan, Ningxia
  - Tangdu Hospital of the Fourth Military Medical University, Xi'an, Shaanxi
  - Qilu Hospital, Jinan, Shandong
  - Jinan Central Hospital, Jinan, Shandong
  - Affiliated Cancer Hospital of Shandong First Medical University, Jinan, Shandong
  - ZhongShan Hospital, Shanghai, Shanghai Municipality
  - The Third Affiliated Hospital of Naval Medical University, Shanghai, Shanghai Municipality
  - Sichuan Cancer Hospital, Chengdu, Sichuan
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Tianjin Cancer Hospital, Tianjin, Tianjin Municipality
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - Shulan（Hangzhou） Hospital, Hangzhou, Zhejiang
  - The First Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang